CLINICAL TRIAL: NCT06280534
Title: Randomized, Double-blind, Single Center Phase Ia Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Food Effects of Single and Multiple Doses of XT1061 in Healthy Subjects
Brief Title: Safety, Tolerability Phase Ia Study of XT1061 in Single and Multiple Doses in Healthy Subjects
Acronym: XT1061
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: XT1061-2022-01
Record Dates: First submitted 2024-01-10; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose group (Experimental): Single doses of 12.5mg (Group 1), 25mg (Group 2), 37.5mg (Group 3), 62.5mg (Group 4, Group A), 125mg (Group 5), 250mg (Group 6), alternative groups (Groups 7-10, 400-800mg).
  Interventions: Drug: Test drug XT1061 capsules and placebo,Single dose group
- Multiple dosing group (Experimental): Multiple administrations of 125mg, 250mg (groups 11, 12) Select one or both groups.
  Interventions: Drug: Test drug XT1061 capsules and placebo，Multiple dosing group
- Food Impact Group (Experimental): 62.5 mg (i.e., single dose Group 4)
  Interventions: Drug: Test drug XT1061 capsules and placebo，Food Impact Group

INTERVENTIONS:
Drug: Test drug XT1061 capsules and placebo,Single dose group — Eight people took capsules of the test drug XT1061 and two people took a placebo.
  Arms: Single dose group
Drug: Test drug XT1061 capsules and placebo，Multiple dosing group — D1-D7 were administered under fasting conditions for 7 consecutive days, of which D1-D6 were administered BID and D7 was administered once in the morning under fasting conditions only.Eight people took capsules of the test drug XT1061 and two people took a placebo.
  Arms: Multiple dosing group
Drug: Test drug XT1061 capsules and placebo，Food Impact Group — Eight people in group A took the test drug XT1061 capsules and two people took placebo, and all eight people in group B took the test drug XT1061 capsules.
  Arms: Food Impact Group

SUMMARY:
A Randomized, Double-Blind, Single-Center Phase Ia Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effects of Single and Multiple Doses of XT1061 in Healthy Subjects.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, dose-escalation, placebo-controlled, single-center clinical study designed to evaluate the safety, tolerability, pharmacokinetic profile and metabolic conversion of XT1061 in healthy subjects with single and multiple administrations, as well as a study of the effect of food on pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign the informed consent before the trial, and fully understand the content, process and possible adverse effects of the trial;
2. They are able to complete the study according to the requirements of the trial protocol;
3. Subjects (including partners) are willing to have no pregnancy plan and voluntarily use effective contraceptive measures within 6 months from screening to the last dose of study drug;
4. Male and female subjects between the ages of 18 and 65 (including borderline values);
5. Male subjects weighing not less than 50 kg and female subjects weighing not less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), BMI within the range of 18-28 kg/m2 (including the threshold value);
6. Physical examination and vital signs are normal or abnormal without clinical significance.

Exclusion Criteria:

1. Allergy (multiple drug and food allergies);
2. Those who smoked more than 5 cigarettes per day in the 3 months prior to the test;
3. History of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
4. Blood donation or significant blood loss (> 450 mL) within three months prior to taking study drug;
5. taking any prescription drug, over-the-counter drug, any vitamin product, herbal remedy, or alcohol within 14 days prior to taking study drug;
6. have taken a special diet (e.g., grapefruit, mango, dragon fruit, grape juice, orange juice, etc., rich in flavonoids or citrus glycosides), or have had strenuous physical activity, or any other factor that affects the absorption, distribution, metabolism, or excretion of the drug within 2 weeks prior to administration of the study drug;
7. Those who have recently made significant changes in their dietary or exercise habits;
8. have taken the study drug, or participated in a clinical trial of the drug within three months prior to taking the study drug;
9. have dysphagia or a history of any gastrointestinal disorder that interferes with the absorption of the drug within 6 months prior to the trial;
10. have any condition that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastroduodenal ulcers
11. clinically significant ECG abnormalities; QTcF >470ms (QTcF=QT/(RR)^0.33); and
12. Female subjects who are breastfeeding or recently preparing for pregnancy or have a positive serum pregnancy result during the screening period or during the course of the trial;
13. Abnormal and clinically significant clinical laboratory tests, or other clinical findings within the 12 months prior to screening that indicate clinically significant disease of the following (including, but not limited to, gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular disease);
14. Positive screening for any of the Hepatitis B Surface Antigen, Hepatitis C Antibody/Hepatitis C Core Antigen, HIV Antigen/Antibody, or Syphilis Spirochete Antibody;
15. Acute illness or concomitant medication from the screening phase until study drug administration;
16. ingestion of chocolate, any caffeinated or xanthine-containing food or beverage 24 hours prior to study drug administration;
17. A positive urine drug screen or a history of substance abuse or drug use within the past five years;
18. serum creatinine clearance ≤ 70 mL/min [formula: Ccr: (140 - age) × body weight (kg) / (0.818 × Scr) (μmol/L), female × 0.85].
19. Those who have special dietary requirements and cannot eat the entire test meal. Or those who did not agree to comply with the drinking arrangements and postural restrictions during the trial;
20. Subjects who, in the opinion of the investigator, have other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | Day 7
  Number of participants who experienced treatment-related adverse events as assessed by CTCAE v5.0.
Cmax | Day 4
  Cmax
Tmax | Day 4
  Tmax
t1/2 | Day 4
  t1/2
AUC | Day 4
  AUC
CL/F | Day 4
  CL/F
Vz/F | Day 4
  Vz/F
CLr/F | Day 4
  CLr/F

SECONDARY OUTCOMES:
Ae0-72 h | Day 4
  Ae0-72 h
Fe0-72 h | Day 4
  Fe0-72 h
bioavailability | Day 4
  geometric mean value ratio

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China